CLINICAL TRIAL: NCT06243965
Title: Is Desmoplastic Stromal Reaction Useful to Modulate Lymph Node Dissection in Sporadic Medullary Thyroid Carcinoma?
Acronym: DSR-MTC
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5547
Record Dates: First submitted 2024-01-15; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Medullary Thyroid Cancer; Medullary Carcinoma; Medullary Tumor; Medullary Neoplasms; Desmoplasia; Desmoplastic; Desmoplastic Reaction; Lymph Node Metastasis; Lymph Node Disease
Keywords: medullary thryoid carcinoma; desmoplasia; lateral neck dissection
MeSH Terms: conditions — Carcinoma, Medullary; Brain Stem Neoplasms; Fibrosis; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The oncologic benefit of lateral neck dissection (LND) during index operation for sporadic medullary thyroid carcinoma (MTC) basing on basal calcitonin (bCT) levels has been questioned due to the potential post-operative complications. This study aims to evaluate desmoplastic reaction (DSR), as predictor of nodal metastases, for definition of surgical strategy.

Data from pathological report of MTC after operations between 1997 and 2022 were collected. The primary endpoint of the study was evaluating the risk factors for nodal metastases. The secondary endpoints analyzed the correlations between DSR and nodal metastases and the sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of DSR for nodal metastases.

DETAILED DESCRIPTION:
Medullary thyroid carcinoma (MTC) is a rare neuroendocrine tumor associated with aggressive biological behavior and a tendency for earlier lymphatic spread compared with differentiated thyroid carcinoma. Most MTCs are sporadic (75%), although some (25%) are hereditary, either familial or occurring in association with multiple endocrine neoplasia type 2 (MEN 2) syndrome. In contrast to hereditary MTC, sporadic MTC presents as multifocal disease only in 10% of patients.

As the most common clinical presentation is an asymptomatic solitary thyroid nodule, sporadic MTC detection is often late. Consequently, it is usually diagnosed as advanced disease, with cervical node involvement in most patients (70%) and compressive symptoms of the upper aerodigestive tract (15% of cases). Indeed, at the time of diagnosis, MTC presents with nodal involvement of central and lateral compartment in 50-81% and 34-81% of patients, respectively. Approximately 5% to 10% of patients with sporadic MTC even present with distant metastasis to the liver, lung, bones, brain and skin.

Complete surgical resection of the primary tumor and regional metastases is the cornerstone for locoregional disease control, since adjuvant therapy remains ineffective for the treatment of sporadic MTC. Moreover, as the number of positive lymph nodes and involved anatomical compartments are cancer-specific prognostic factors, early and accurate diagnosis of regional lymph nodes involvement is crucial for determining the surgical strategy. However, pre-operative diagnosis of MTC-related nodal disease is challenging due to the low sensitivity of imaging studies on detecting regional spread. Therefore, clinical decisions are often based upon biomarkers, mainly basal calcitonin levels, to predict nodal involvement and plan the surgical extent. Several associations have advocated in favor of this approach, although not with a strong recommendation, by suggesting prophylactic neck dissections based on basal calcitonin levels, especially for the lateral compartments. However, recent studies challenge this approach since a significant portion of patients were exposed to operations with increased morbidity without nodal spread on final histology or obvious survival benefits. As a consequence, the need to develop new predictive tools to tailor the surgical extent to each patient is paramount.

Desmoplasia, defined as the newly paraneoplastic formed stromal reaction surrounding the invasive epithelial tumor cells, has recently resurfaced as a morphological parameter with distinct clinical relevance in MTC. Significant correlation of desmoplasia with lymph node metastasis has been described in literature, with a higher specificity in predicting the nodal metastasizing pattern when compared with other morphological features. More specifically, the absence of desmoplasia on frozen section and definitive histopathology has been strongly associated with the absence of nodal metastases. As such, desmoplasia may have a crucial role in guiding surgical extent in the future.

The aim of this study is to evaluate the correlation between desmoplasia and nodal involvement in unifocal sporadic MTC in our experience.

ELIGIBILITY:
Inclusion Criteria:

* All adults patients who underwent index procedure for sporadic unifocal MTC whose specimens were retrospectively re-evaluated by an expert endocrine pathologist (E.D.R.) for DSR were candidates for inclusion.

Exclusion Criteria:

* hereditary MTC
* sporadic multifocal MTC
* index operation in another center
* incidental diagnosis of MCT after less than total thyroidectomy and bilateral central neck dissection
* less than 6-months-follow-up
* patients < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults patients who underwent index procedure between January 1997 and December 2022 in our center for sporadic unifocal MTC whose specimens were retrospectively re-evaluated by an expert endocrine pathologist (E.D.R.) for DSR were candidates for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 1997-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Risk factors for nodal metastases | January 1997-December 2022
  The primary endpoint of the study consists in the evaluation of risk factors for nodal metastases in patients with histopathologic report of medullary thryoid carcinoma

SECONDARY OUTCOMES:
Correlations between desmoplastic stromal reaction and nodal metastases | January 1997-December 2022
  The secondary endpoints consist in the evaluation of correlations between desmoplastic stromal reaction and nodal metastases and in the sensitivity, specificity, PPV and PNV of desmoplastic stromal reaction for nodal metastases in patients with histopathologic report of medullary thyroid carcinoma

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Reasonable requests will be evaluated by the Principal Investigator of our study